CLINICAL TRIAL: NCT05379673
Title: Recovery of Ventilation After General Anesthesia for Robotic-Assisted Laparoscopic Nephrectomy or Prostatectomy: The Effect of Oxygen Supplementation
Brief Title: The Effect of Hyperoxia on Ventilation During Recovery From General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, Professor, Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-63878
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ventilatory Depression; Postoperative Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: In the post-anesthesia care unit (PACU), participants will be randomized to receive conservative (titrated to an SpO2 between 90 and 94%) versus liberal (titrated to SpO2 > 96%) oxygen supplementation, via a non-rebreather mask.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the received treatment. The investigators, who will monitor the patients and collect the data in the PACU, will be blinded to the primary outcome, but not to the received treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- "Conservative O2 Supplementation" (Active Comparator): Oxygen administration will be titrated to a oxyhemoglobin saturation (SpO2) between 90 and 94%.
  Interventions: Other: Oxygen Gas for Inhalation
- "Liberal O2 Supplementation" (Experimental): Oxygen administration will be titrated to an SpO2 > 96%.
  Interventions: Other: Oxygen Gas for Inhalation

INTERVENTIONS:
Other: Oxygen Gas for Inhalation — Oxyhemoglobin saturation (SpO2) higher than 96% vs SpO2 between 90% and 94%.

SUMMARY:
In this randomized-controlled trial the investigators will examine the effect of oxygen supplementation on the recovery of breathing for 90 minutes in the immediate post-anesthesia period starting from extubation of the trachea.

DETAILED DESCRIPTION:
In a pilot randomized-controlled trial (NCT04723433) the investigators found that hyperoxia, compared with standard O2 supplementation, enhanced ventilation, as estimated by the fraction of time at a transcutaneous PCO2 (TcPCO2) > 45 mmHg.

More specifically, patients treated with hyperoxia (O2 titrated to: SpO2 > 96%, N=10; Liberal O2) for 90 minutes post-anesthesia, spent 61.2% of the time at TcPCO2 > 45 mmHg, compared with 80.6% of the time in those receiving standard O2 supplementation (O2 titrated to: SpO2 between 90-94%, N=9; Conservative O2 - between-group difference of 19.4% (95% CI: -18.7% to 57.6%), ANCOVA adjusted P = 0.140]. Results were consistent across the 90-min monitoring period. With an observed effect size of 0.73, it was estimated that 30 participants per group are required, to demonstrate this difference with a power of 80% at a two-sided alpha of 5%.

In the present confirmative randomized controlled trial, the investigators plan to estimate and compare the cumulative segment of time during which the transcutaneous partial pressure of carbon dioxide will exceed an upper limit of 45 mmHg (i.e., TcPCO2 > 45 mmHg) for the 90-min-long post-anesthesia period, between the conventional (titrated to an oxygen saturation > 96%) and the conservative (titrated to O2 saturation 90-94%) O2 supplementation interventions.

Hypothesis: Conservative use of O2 (titrated to an SpO2: 90 - 94%), will be associated with more hypoventilation (i.e., more time spent with an TcPCO2 > 45 mmHg) during recovery from general anesthesia, compared to liberal O2 supplementation (SpO2 > 96%).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Body mass index (BMI) less than 40 kg/m2
* Scheduled to undergo robotic-assisted radical laparoscopic nephrectomy or prostatectomy.

Exclusion Criteria:

* Patients with a diagnosis of chronic obstructive pulmonary disorder (COPD), severe neurological, cardiopulmonary, psychiatric, or untreated thyroid disorder
* Chronic pain condition that is being treated with opioids
* Patients with a hematocrit lower than 30% at the end of surgery, or those with an excessive blood loss, requiring transfusion of blood products during surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous partial pressure of carbon dioxide (TcPCO2) | Ninety -minute period beginning immediately post-anesthesia.
  The cumulative segment of time during which the transcutaneous partial pressure of carbon dioxide (TcPCO2: primary outcome) will exceed an upper limit of 45 mmHg (i.e., TcPCO2 > 45 mmHg)

SECONDARY OUTCOMES:
Apnea / hypopnea index (AHI) | Ninety -minute period beginning immediately post-anesthesia.
  The number of apnea /hypopnea episodes detected using respiratory inductance plethysmography and nasal pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, MD, PhD, Principal Investigator — Professor, Department of Anesthesiology, Stanford University Medical School
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No